CLINICAL TRIAL: NCT04604600
Title: Multimodal Biomarkers for Diagnosis and Prognosis in Vascular Cognitive Impairment
Brief Title: Multimodal Biomarkers for Diagnosis and Prognosis in VCI
Acronym: VCI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201912098MINB
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Vascular Cognitive Impairment; Alzheimer Disease
Keywords: Vascular Cognitive Impairment; ApoE genotype; Amyloid PET; Brain MRI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amyloid PET、T807 PET (Experimental): PET/CT
  Interventions: Drug: amyloid PET

INTERVENTIONS:
Drug: amyloid PET — Dynamic PET acquisition for 70 minutes will be acquired after injection of 10±5 mCi 11C-PiB.

SUMMARY:
We will try to

1. establish the correlation of plasma Aβ40 and Aβ42 level, ApoE genotype, MRI imaging markers in the diagnosis and prognosis of VCI patients
2. understand more on the pathophysiology of VCI.

DETAILED DESCRIPTION:
Background and objectives Owing to the aging problem, cognitive impairment has been a worldwide health issue. Vascular cognitive impairment (VCI) and Alzheimer's disease (AD) are the two most common causes. It has been reported that VCI and AD share many common risk factors. MRI is essential in assessing the extent, location and type of vascular lesions. Amyloid PET has been used in detecting cerebral amyloid burden non-invasively since 2004. There are only small number of studies using amyloid PET in VCI and the results are still controversial. In the current proposal, we will investigate

1. the correlation of clinical risk factors, ApoE genotype, various MRI markers, and amyloid PET expression
2. assess the influence of ApoE genotype on different biomarkers, including MRI markers, amyloid retention, and plasma Aβ40 and Aβ42 levels
3. the potential of amyloid PET as a prognostic factor for VCI patients.

Materials and methods This study will be conducted in National Taiwan University Hospital and Bei-Hu Branch Hospital. Sixty clinical diagnosed VCI, 30 AD patients and 30 normal subjects will be enrolled in this 3-year prospective study. We will collect vascular risk factors, neuropsychological tests, 10 cc venous blood for plasma Aβ40, Aβ42, total tau and phosphorylated level measurement by IMR assay, ApoE genotype, brain MRI, and amyloid PET of each patient and control subject. All the data will be analyzed together.

Expected Results We will try to

1. establish the correlation of plasma Aβ40 and Aβ42 level, ApoE genotype, MRI imaging markers in the diagnosis and prognosis of VCI patients
2. understand more on the pathophysiology of VCI.

ELIGIBILITY:
Inclusion Criteria:

-

I. Vascular cognitive impairment patients:

1. Age older than 20 years.
2. Clinical diagnosis:

   1. At least one obstacle to executive function, attention, memory, language and visual space function.
   2. Affected activities of daily living.
   3. Brain MRI showing cerebrovascular disease.
3. Patient agrees to participate in the study and is willing to receive 11C-PiB PET.

II. Alzheimer's disease (AD) patients:

1. Age older than 20 years.
2. Clinical diagnosis:

   1. Amnesia or non-amnesia (language, visual space, executive ability) performance.
   2. Affected activities of daily living.
3. Patient agrees to participate in the study and is willing to receive 11C-PiB PET.

III. Normal controls:

1. Age older than 20 years.
2. No neurological or psychiatric history.
3. Patient agrees to participate in the study and is willing to receive 11C-PiB PET.

Exclusion Criteria:

-

I. Vascular cognitive impairment patients:

1. Have other illnesses, including people with drug / alcohol abuse / addictivity within three months.
2. Patient cannot accept brain magnetic resonance imaging or 11C-PiB PET, such as agitation and inability to cooperate, allergy to contrast agents, hemodynamic instability (blood pressure, pulse, or blood oxygen is not in the normal range), and a heart rhythm regulator has been implanted , Have ever undergone intracranial aneurysm clamp surgery, claustrophobia and hemodynamic instability.
3. Pregnant woman or intends to be pregnant in the near future.
4. Patient who is breast feeding or intends to.
5. Allergic to 11C-PiB, or with severe drug allergy history.
6. Patient or the family refuses to participate in the study.

II. Alzheimer's disease (AD) patients:

1. Have other illnesses, including:

   1. Cognitive disorders caused by cerebrovascular diseases (the decline in cognitive function is closely related to the time of stroke, multiple large-scale necrosis, and severe white matter lesions).
   2. The main manifestation of dementia is Lewy body dementia
   3. Symptoms are behavioral variation of frontotemporal dementia.
   4. The symptoms are obviously semantic progressive aphasia.
   5. Symptoms are not fluent in primary progressive aphasia.
   6. Other comorbidities that affect cognitive function (including other active neurological diseases, or non-neurological diseases but the disease or the treatment used will affect cognitive function)
2. Patient cannot accept brain magnetic resonance imaging or 11C-PiB PET, such as agitation and inability to cooperate, allergy to contrast agents, hemodynamic instability (blood pressure, pulse, or blood oxygen is not in the normal range), and a heart rhythm regulator has been implanted , Have ever undergone intracranial aneurysm clamp surgery, claustrophobia and hemodynamic instability.
3. Pregnant woman or intends to be pregnant in the near future.
4. Patient who is breast feeding or intends to.
5. Allergic to 11C-PiB, or with severe drug allergy history.
6. Patient or the family refuses to participate in the study.

III. Normal controls:

1. Patient cannot accept brain magnetic resonance imaging or 11C-PiB PET, such as agitation and inability to cooperate, allergy to contrast agents, hemodynamic instability (blood pressure, pulse, or blood oxygen is not in the normal range), and a heart rhythm regulator has been implanted , Have ever undergone intracranial aneurysm clamp surgery, claustrophobia and hemodynamic instability.
2. Pregnant woman or intends to be pregnant in the near future.
3. Patient who is breast feeding or intends to.
4. Allergic to 11C-PiB, or with severe drug allergy history.
5. Patient or the family refuses to participate in the study.
6. high risk as assessed by a doctor.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
PET imaging | in 3 days
  PET data will reconstruct with ordered set expectation maximization, corrected for attenuation, and each frame will be evaluated to verify adequate count statistics and absence of head motion.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No